CLINICAL TRIAL: NCT03082807
Title: Investigating the Effects of Negative Calorie Diet Compared With Low-calorie Diet Under Exercise Condition on Weight Loss and Lipid Profile in Overweight/Obese Middle-aged and Older Men
Brief Title: Dietary Guide in Active Older Adult Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P.L.Shupik National Medical Academy of Post-Graduate Education (Other)
Responsible Party: Principal Investigator, Mohammadreza Rezaeipour, MD, PhD, Asst. Prof. of sports medicine (sports injury and corrective movement), University of Sistan and Baluchestan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: no Grant 6
Record Dates: First submitted 2017-03-07; First posted 2017-03-17 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Men; Diet Modification; Obesity; Overweight; Life Style; Weight Loss
Keywords: Caloric Restriction; Diet; Exercise; Obesity; Overweight; Sedentary lifestyle; weight loss; Men
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Obesity; Overweight; Weight Loss; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group I (Experimental): Study group I (18 participants) received the NCD with exercise (NCDsport). This groups had 5% caloric restriction from their maintenance energy requirements and 10% increase in energy expenditure through structured regular exercise.
  Interventions: Dietary Supplement: NCDsport
- Study group II (Experimental): Study group II (19 participants) received the low-calorie diet with exercise (LCDsport). This groups had 5% caloric restriction from their maintenance energy requirements and 10% increase in energy expenditure through structured regular exercise.
  Interventions: Dietary Supplement: LCDsport

INTERVENTIONS:
Dietary Supplement: NCDsport — Negative Calorie Diet supplemented with exercise
  Other Names: group I
  Arms: Study group I
Dietary Supplement: LCDsport — Low-Calorie diet with exercise
  Other Names: group II
  Arms: Study group II

SUMMARY:
The present study aimed to determine the effects of negative-calorie diet supplemented with exercise, on weight loss and lipid profile, and to compare its efficiency with low-calorie diet with exercise among elderly adult men with abnormal weight gain.

DETAILED DESCRIPTION:
Background and Aim: Negative-calorie diet is among the popular dieting guides for weight loss; however, there is still little knowledge about this method. The present study aimed to determine the effects of negative-calorie diet supplemented with exercise, on weight loss and lipid profile, and to compare its efficiency with low-calorie diet with exercise among elderly adult men with abnormal weight gain.

Materials and Methods: Participants included sedentary men (age 45-75 years) with overweight or obesity (n=37). They were randomly divided into 2 groups including negative calorie diet with exercise, and low-calorie diet with exercise. Of all 37 participants, 30 persons completed the treatment. The weight assessment parameters including change in weight and body composition, blood sample tests were performed pre- and three month post-intervention.

ELIGIBILITY:
Inclusion Criteria:

Non-smokers and weight-stable (± 2 kg, for more than one year) with no history of regular exercise in at least three months before the study.

Exclusion Criteria:

History of CVD and other disorders such as diabetes, depression, eating disorders, chronic medications, kidney disease, cancer, food allergies or intolerances to items used in meals. Subjects with abnormality in thyroid or Electrocardiograph, any history of anti-obesity medication or weight loss drugs or dietary supplementations for weight control.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants were non-smokers and weight-stable (± 2 kg, for more than one year) with no history of regular exercise in at least three months before the study.
Enrollment: 37 (Actual)
Dates: Start 2011-02-25 (Actual); Primary Completion 2012-09-20 (Actual); Study Completion 2012-12-15 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline
  assessed in kg
Total cholesterol (Total-C) | Baseline
  assessed in mg/dl
High-density lipoprotein -cholesterol (HDL-C) | Baseline
  assessed in mg/dl
Low-density lipoprotein -cholesterol (LDL-C) | Baseline
  assessed in mg/dl
Triglycerides (TG) | Baseline
  assessed in mg/dl

SECONDARY OUTCOMES:
Weight | 3-month
  assessed in kg
Total cholesterol (Total-C) | 3-month
  assessed in mg/dl
High-density lipoprotein -cholesterol (HDL-C) | 3-month
  assessed in mg/dl
Low-density lipoprotein -cholesterol (LDL-C) | 3-month
  assessed in mg/dl